CLINICAL TRIAL: NCT03932214
Title: Infrared Illumination for Difficult Peripheral Venous Catheterization in Adult Critically-ill Patients
Brief Title: Infrared for Peripheral Venous Catheterization in the Critically-ill
Acronym: ICARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRIP-18-0617
Record Dates: First submitted 2019-04-26; First posted 2019-04-30 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Venous Catheterization
Keywords: venous access; illumination, infrared; critically-ill; catheterization
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Subjects will be divided into two groups with a 1: 1 ratio. Each patient will be assigned to one of the following 2 arms:
  - Usual technique : Visualization of the vein to be catheterized will be done directly. without infrared illumination.
  or
  -Use of the Accuvein® device: Visualization of the vein to be catheterized will be done with infrared illumination.
  In both groups, catheterization will be carried out according to the usual technique in accordance with the recommendations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infrared illumination group (Experimental): The nurse uses the Accuvein® device to identify the veins before puncture.
  Interventions: Device: ACCUVEIN
- Control group (No Intervention): The nurse proceeds as usual (visual identification in the light of the room and palpation)

INTERVENTIONS:
Device: ACCUVEIN — The nurse uses the Accuvein® device to identify the veins before puncture and then proceeds as usual, under illumination of the device.
  Arms: Infrared illumination group

SUMMARY:
Peripheral venous catheterization is a fundamental part of the management of critically-ill patients, especially for administration of intravenous emergency treatments. In general, it is preferred to central catheterization whenever possible, since it is less invasive, achievable immediately by the nurse, and responsible for fewer complications.

Venous access difficulties are frequent in critically-ill patients. Among tools proposed to improve the practice of peripheral catheterization, ultrasound and infrared illumination are the most studied, the latter being simpler. Infrared illumination has never been evaluated in intensive care. However, the delay or failure of peripheral catheterization is highly detrimental in the context of resuscitation as it may delay or impede appropriate management of vital emergencies. Our study will focus on the peripheral venous catheterization of the upper limbs, as these are the reference site for this technique The objective is to evaluate the interest of infrared illumination (AccuVein AV500®) for the primary success (first puncture) of peripheral venous catheterization of the upper limbs in patients with resuscitation at risk of catheterization venous difficult.

It is a comparative, superiority, prospective, multicenter, randomized, controlled, open-label, phase III trial. Subjects will be divided into two groups with a 1: 1 ratio. Nurses at participating centers will be trained for the use of the device prior to the start of the study; the use of the device is singularly easy and intuitive.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years; Hospitalization in intensive care;
* Need for a peripheral venous catheter;
* Risk of difficult peripheral venous catheterization. In practice, this risk will be considered present if it is impossible to palpate and / or visualize the upper end of the target vein and / or if the estimated vein diameter is smaller than 2mm. This definition is derived from the A-DIVA score (Loon FAJ van et al3).
* Affiliation to the social security

Exclusion Criteria:

* Patient who has already been enrolled in the ICARE study during the current hospitalization;
* Refusal of patient's participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of primary success of peripheral venous catheterization in the upper limbs. | Day 1
  success defined as the need of a single puncture for the effective catheterization.
  The effective catheterization is confirmed by obtaining venous reflux by declivity of the infusion bag.

SECONDARY OUTCOMES:
Number of punctures required for peripheral venous catheterization. | Day 1
Rate of failure of the procedure, defined by the absence of placement of a peripheral venous catheter before the end of the procedure | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Fabien BOUSSELY, senior officer, Principal Investigator — Assistance publique des hopitaux de Paris
Locations (1):
- Henri-Mondor Hospital, Créteil, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION

REFERENCES:
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Loon FHJV, Puijn LAPM, Houterman S, Bouwman ARA. Development of the A-DIVA Scale: A Clinical Predictive Scale to Identify Difficult Intravenous Access in Adult Patients Based on Clinical Observations. Medicine (Baltimore). 2016 Apr;95(16):e3428. doi: 10.1097/MD.0000000000003428. PMID 27100437
- [Derived] Ouedraogo R, Alves A, Bruant A, Sy O, Tabra Osorio C, Schortgen F, Chenal A, Contou D, Krzyzaniak L, Fartoukh M, Le Joncour M, Mongardon N, Ait Benaissa L, Da Silva D, Bouguerra M, Demeret S, Tanguy Dubois S, Starczala E, Petyt C, Schmidt M, Dezellus S, Georger JF, Pallud AC, Carras D, Boussely F, Audureau E, Mekontso Dessap A. Infrared illumination for difficult peripheral venous catheterisation in critically ill adult patients: the prospective, randomised, multicentre ICARE trial. BMJ Open. 2025 Feb 6;15(2):e090611. doi: 10.1136/bmjopen-2024-090611. PMID 39915026